CLINICAL TRIAL: NCT00449527
Title: A Two-week, Randomised, Double-blind Study Assessing the Onset of Effect Questionnaire Administered Daily Versus Weekly in Adult Subjects (≥ 18 Years) With Mild to Moderate Asthma, Receiving SYMBICORT® pMDI 80/4.5 μg x 2 Actuations Twice Daily or Budesonide HFA pMDI 80 μg x 2 Actuations Twice Daily
Brief Title: A Two-week Study Assessing the Onset of Effect Questionnaire (OEQ) Administered Daily Versus Weekly in Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5896C00023
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Mild asthma; Moderate asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Budesonide/formoterol pMDI
  Other Names: Symbicort
Drug: Budesonide HFA pMDI

SUMMARY:
The purpose of this study is to demonstrate whether subjects respond similarly to the Onset of Effect Questionnaire (OEQ) using a 1 week recall period versus a 1 day recall period.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, > 18 years of age
* Mild to moderate asthma requiring treatment with an inhaled corticosteroid
* Diagnosis of asthma for at least 6 months

Exclusion Criteria:

* Subjects requiring treatment with systemic corticosteroids (e.g., oral, parenteral, ocular)
* Subjects with severe asthma, as judged by investigator
* Any significant disease or disorder that may jeopardize a subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2007-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate whether subjects respond similarly to the Onset of Effect Questionnaire (OEQ) items 2 and 5 using a 1 week recall period versus a 1 day recall period.

SECONDARY OUTCOMES:
To demonstrate the value to subjects of feeling an asthma maintenance medication begins to work right away; to assess the correlation between subject's responses to weekly/daily Onset of Effect Questionnaires with lung function and with diary variables.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas LG Andersson, MD, Study Director — AstraZeneca
Locations (44):
- United States (44):
  - Research Site, Tuscumbia, Alabama
  - Research Site, Fort Smith, Arkansas
  - Research Site, Long Beach, California
  - Research Site, Orange, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Valrico, Florida
  - Research Site, River Forest, Illinois
  - Research Site, Council Bluffs, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Bowling Green, Kentucky
  - Research Site, Florence, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, City of Saint Peters, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Papillion, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Skillman, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, North Syracuse, New York
  - Research Site, Rochester, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Collegeville, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, South Burlington, Vermont
  - Research Site, Bellingham, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington

REFERENCES:
- [Derived] Leidy NK, Gutierrez B, Lampl K, Uryniak T, O'Brien CD. Can patients with asthma feel inhaler therapy working right away? Two clinical trials testing the effect of timing of assessment on patient perception. J Asthma. 2009 Dec;46(10):1006-12. doi: 10.3109/02770900903301260. PMID 19995138
- See also: Related Info — http://www.asthmaclinicaltrials.com